CLINICAL TRIAL: NCT05783180
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ (Liposomal Bovine Lactoferrin (LbLf) and Liposomal Zn (LZn)) and Standard of Care (SOC) vs SOC in the Treatment of Non-hospitalized Patients With COVID-19
Brief Title: LACTYFERRIN™ Forte and ZINC Defense™ and Standard of Care (SOC) vs SOC in the Treatment of Non-hospitalized Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided not to move forward with the trial
Sponsor: Jose David Suarez, MD (Other)
Collaborators: Sesderma S.L. (Unknown); Westchester General Hospital Inc. DBA Keralty Hospital Miami (Unknown); MGM Technology Corp (Unknown)
Responsible Party: Sponsor-Investigator, Jose David Suarez, MD, Principal investigator, Keralty Hospital, Miami
Organization: Keralty Hospital, Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SES-LFZN-001
Record Dates: First submitted 2023-03-09; First posted 2023-03-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: Liposomal lactoferrin; liposomal Zinc; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Treatment Group: Sesderma LACTYFERRIN™ Forte (64mg/20ml, TID) and Sesderma ZINC Defense™ (20mg/20ml QD) + SOC (N=20).
  Control group: Placebo +SOC (N=20) Intervention groups At baseline, subjects will be randomized in a 1:1 ratio to either treatment or control groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two teams will be involved in the trial unblinded team that will randomized the subjects and dispense the investigational product and the blinded team that will be involved in the clinical evaluations and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Sesderma LACTYFERRIN™ Forte (64mg/20ml, TID) and Sesderma ZINC Defense™ (20mg/20ml QD) + SOC (N=20).
  Interventions: Drug: Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™
- Control (Placebo Comparator): Placebo +SOC (N=20)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ — Sesderma LACTYFERRIN™ Forte (64mg/20ml, TID) and Sesderma ZINC Defense™ (20mg/20ml QD)
  Arms: Treatment
Drug: Placebo — Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ (Placebo)
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn about the safety and efficacy of Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ in non-hospitalized patients with COVID-19.

The main question is:

Is there a reduction in the signs and symptoms of COVID-19 from baseline to end of treatment? Participants will complete the following activities.

* Screening and first day of treatment
* Treatment that will be administered for up to 10 days, two treatment evaluation visits will be completed
* After treatment completion. Two visits are scheduled, one 28 days after the last dose and the other 60 days after the last dose.

Researchers will compare Treatment Group (Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ + Standard of care (SOC)) with the Control group (Placebo +SOC) to see if there is Reduction in the signs and symptoms of COVID-19 at the end of treatment

DETAILED DESCRIPTION:
This is a placebo-controlled, randomized, parallel-group, adaptive, phase 2 study to evaluate the safety and efficacy of Sesderma LACTYFERRIN™ Forte and Sesderma ZINC Defense™ (LbLf+LZn) + SOC compared to Placebo+SOC in non-hospitalized patients with COVID-19. The primary endpoint is the reduction in the signs and symptoms of COVID-19 from baseline to D11/D28 (end of treatment).

The study duration will be up to 70 days including.

* Screening and randomization (Day0/D1): Screening and the first day of treatment
* Treatment period: from (D0 to D10). Treatment will be administered for up to 10 days, and treatment evaluation visits on D11 (EOT) and D28.
* Follow-up (FU): Will start after treatment completion on day 10. Two visits are scheduled during this period: one 28 days after the last dose (D38) and the other 60 days after the last dose (D70).

Patient population None hospitalized Individuals with mild to moderate SARS-CoV-2 infection with less than 7 days of symptoms evolution. This corresponds to a score of 1 or 2 (moderate to mild disease) on the WHO 9-point ordinal scale

Number of subjects Approximately: 40

Treatment Group: Sesderma LACTYFERRIN™ Forte (64mg/20ml, TID) and Sesderma ZINC Defense™ (20mg/20ml QD) + SOC (N=20).

Control group: Placebo +SOC (N=20)

Intervention groups At baseline, subjects will be randomized in a 1:1 ratio to either treatment or control groups.

ELIGIBILITY:
INCLUSION CRITERIA

* Patient or legally authorized representative must be willing to sign an informed consent.
* Male or female ≥18 years of age at the time of enrollment.
* COVID-19 diagnosis confirmed by SARS-CoV-2 detection by polymerase chain reaction (PCR) or other commercial or public health assays in any specimen documented by any of the following:
* PCR positive in samples collected ≤ 72h.
* PCR positive in samples collected >72h and less than 7 days of disease progression.
* Mild to moderate symptoms of COVID-19 as determined by investigators following the criteria from NIH COVID 19 Treatment Guidelines for (APPENDIX I. SEVERITY OF ILLNESS CATEGORIES).

EXCLUSION CRITERIA

* Hospitalized patients.
* Breast-feeding or pregnant (any woman of childbearing age and potential must have a negative test within 24 hours of starting treatment).
* Allergy to any of the components of the study medication.
* AST or ALT > x3 the upper limit value
* Estimated Glomerular Filtration Rate (eGFR) < 30
* Concomitant antiviral therapy such as lopinavir or ritonavir
* Concomitant immunosuppressive or immunomodulatory drugs (e.g., interleukins, interleukin antagonists or receptor blockers, anticancer drugs, immunosuppressant)
* Concomitant therapy with corticosteroids at a dose > 20mg per day was administered for more than 14 days before the study medication.
* Human immunodeficiency virus infection under highly active antiretroviral therapy (HAART).
* Has participated in another clinical trial within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in the signs and symptoms of COVID-19 from baseline to Day 11 (end of treatment, EOT). | 11 days (one day after last study medication dose)
  The scale used by Serrano et al., 2020 during the Phase 1 Sesderma LACTYFERRIN™ Forte trial quantified the presence of COVID-19 signs and symptoms, and their reduction during treatment time will be used in this phase with the same purpose

SECONDARY OUTCOMES:
The proportion of patients with disease progression on Day 28 | up to 28 days after first study medication dose
  The proportion of patients with disease progression on Day 28, are defined as the proportion of patients who are not alive or who have respiratory failure. Respiratory failure is defined as the need for invasive or non-invasive mechanical ventilation, high-flow oxygen, or ECMO.
Time to recover or Odds of Ratio for Improvement in WHO 9-point ordinal scale | 5,11 and 28 days after first study medication dose
  Time to recover or Odds of Ratio for Improvement in WHO 9-point ordinal scale from Baseline to D5/D11 (EOT)/D28.
The change in blood levels of inflammatory biomarkers | 5,11 and 28 days after first study medication dose
  The change in blood levels CRP, CRP/albumin, ferritin, iron, and D-Dimer from baseline, D5, D11 (EOT), and 28.
Adverse event | through study completion, an average of 70 days
  Assessment of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jose D Suarez, Principal Investigator — Keralty Hospital, Miami
Locations (1):
- Keralty Hospital Miami, Miami, Florida, United States

REFERENCES:
- [Background] Martorell P, Llopis S, Gonzalez N, Ramon D, Serrano G, Torrens A, Serrano JM, Navarro M, Genoves S. A nutritional supplement containing lactoferrin stimulates the immune system, extends lifespan, and reduces amyloid beta peptide toxicity in Caenorhabditis elegans. Food Sci Nutr. 2016 Jul 28;5(2):255-265. doi: 10.1002/fsn3.388. eCollection 2017 Mar. PMID 28265360